CLINICAL TRIAL: NCT01658137
Title: Dietary Intervention Trial to Understand the Mechanism Underlying the 9p21 Variant Interaction With High Fruits and Vegetable Consumption
Brief Title: Diet Intervention and GEnetic STudy (DIGEST-Pilot)
Acronym: DIGEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sonia Anand, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIGEST-Pilot
Record Dates: First submitted 2012-07-28; First posted 2012-08-06 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases; Inflammation; Dyslipidemias; Blood Pressure; Hyperglycemia
Keywords: diet; dietary pattern; gene; gene expression; epigenomics; diet-gene interaction; inflammation; 9p21; fruits; vegetables
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Dyslipidemias; Hyperglycemia | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Typical Western Diet (Active Comparator): The comparator dietary pattern ("Typical Western Diet") approximates the inflammatory dietary pattern typically consumed by North Americans. It contains refined grains, processed foods, dairy fat, meats, sugar and high glycemic index foods, and few fruits, nuts, legumes, and vegetables. The fruits and vegetables are highly processed (e.g. juices) and lower in micronutrients than those in the intervention diet. The saturated fat content of this diet does not meet national guidelines for health. The polyunsaturated fat:saturated fat ratio is ~0.5 (low).
  Interventions: Other: Typical Western Diet
- Prudent Diet (Experimental): The experimental dietary pattern ("Prudent Diet") is based on intakes of foods hypothesized to have beneficial effects on inflammation and long-term health. This dietary pattern includes micronutrient and macronutrient levels consistent with healthy eating in epidemiological studies and randomized controlled trials. The diet is constructed with low-fat dairy products, fish, chicken, and lean meats to minimize saturated fat and increase protein and calcium. The diet is rich in fruits, vegetables, whole grains, nuts, legumes, and seeds that are good sources of potassium, magnesium, and dietary fiber. This diet provides a 'favorable' macronutrient profile that is low in saturated fat, has a polyunsaturated/saturated fat ratio of ~1.0 (high), and low in high glycemic index carbohydrates.
  Interventions: Other: Prudent Diet

INTERVENTIONS:
Other: Prudent Diet — This intervention lasts 2 weeks (14 days).
  Arms: Prudent Diet
Other: Typical Western Diet — This intervention lasts 2 weeks (14 days).
  Arms: Typical Western Diet

SUMMARY:
Genetic factors contribute to risk factors for cardiovascular disease, such as blood lipids, blood pressure, obesity, diabetes, and may also influence dietary choices, physical activity, and responses to stress. The most robust genetic variant associated with myocardial infarction (MI) is the 9p21 variant, which may raise the risk of MI by up to 40% in those who carry 2 copies of the gene. The investigators recently found that among those who carry the 9p21 variant, the risk of MI may be "turned off" if individuals eat a diet high in fruits and vegetables. The investigators seek to determine how a "prudent" or "anti-inflammatory" diet interacts with the 9p21 risk allele to alter the risk of MI.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death globally. The majority of CVD is explained by conventional risk factors including cigarette smoking, abnormal lipids, high blood pressure, obesity, diabetes, and health behaviours including dietary intake, physical activity, and psychosocial stressors. Genetic factors contribute to the development of these risk factors, and directly to CVD through other novel pathways. Since the advent of high throughput chip-based genotyping, more than 30 genetic variants have been found to be associated with myocardial infarction. The most robust genetic variant which has been consistently associated with myocardial infarction and other forms of arterial disease is the 9p21 variant. This genetic variant located on Chromosome 9 is common in the population, with 50% of people carrying one copy of the risk allele, and an additional 25% of the population carrying two copies of the risk allele. Compared with those with no copies of the risk allele, the risk of myocardial infarction with one copy of the risk allele is 15-20% higher, and the increased risk among carriers of 2 risk alleles is 20-40%. To date the exact mechanism by which the 9p21 variant increases the risk of myocardial infarction is unknown, although some data suggests that other genes and pathways associated with cell proliferation and inflammation are involved. Recently we made the observation that among carriers of the 9p21 variant, the risk of MI may be "turned off" if individuals consumed a diet high in fruits and vegetables. However the "mechanism" underlying this interaction is unknown. We seek to discover how a "Prudent" (i.e. anti-inflammatory) diet interacts with the 9p21 risk allele(s) to alter the risk of myocardial infarction.

We postulate that a "Prudent" diet (i.e. a diet high in fruits, vegetables, whole grains, non-processed foods) in comparison to a "Western" or "inflammatory diet" (eg, a typical North American diet high in saturated fats and processed foods) will differentially alter the gene expression (measured by RNA) of the 9p21 locus, change the epigenetic marks in this region, and alter several inflammatory markers suspected to mediate the effect of 9p21 on CVD risk (eg, hs-CRP, IF-alpha21, IFN-γ , interleukin 1-alpha, interleukin 1-beta, and interleukin 6) among people with one or two copies of the risk allele compared to people without the risk allele.

The proposed study offers an unique approach to studying dietary relationships with endpoints believed to be influenced by 9p21 gene variants. Rather than testing nutritional supplements, our results will be generalizable to the setting of most dietary counseling practices, which aim to alter dietary patterns, not specific nutrients. This trial will help us to unravel the basis for gene-diet interactions and gain a greater understanding of how inflammation is linked to the development of atherosclerosis, CVD, and possibly some cancers.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* non-smokers
* Body-Mass-Index <=30 kg/m^2
* willing and able to cook, prepare, and eat provided study foods

Exclusion Criteria:

* Aged below 18 years or above 80 years
* current tobacco smoking
* Body mass index above 30 kg/m2
* Unwillingness or inability to cook, prepare and eat provided study foods (e.g. for medical, philosophical, or religious reasons)
* Excessive use of alcohol (>14 drinks/week in men; >7 drinks/week in women)
* Significant morbidity that would interfere with participation or assessment, including :
* Cancer
* HIV
* chronic renal disease
* renal failure
* Hepatitis/Jaundice
* Liver Disease
* Chronic Obstructive Pulmonary Disease
* Inflammatory bowel disease (Crohn's / Colitis)
* High blood or urine sugar/diabetes
* High blood cholesterol or triglycerides
* Angina/Heart attack/Coronary artery disease
* Heart failure
* Other heart disease
* Angioplasty (balloon opening of an artery) or coronary bypass surgery
* Medications or nutritional supplements (including multivitamins) that could affect outcome measurements. Excluded medications would include:
* Lipid/cholesterol lowering pills
* Insulin/oral hypoglycemic agents
* Medication for stroke
* Antibiotics
* oral contraceptives
* hormone replacement therapy
* non-steroidal anti-inflammatory drugs
* corticosteroids
* unwillingness to stop nutritional supplements 1 week prior to and for duration of intervention
* anticipated difficulties maintaining body weight (e.g. athletic training)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
gene expression measuring ANRIL production | baseline and 2 weeks
epigenetic marks | baseline and 2 weeks

SECONDARY OUTCOMES:
high-sensitivity C-reactive protein | baseline and 2 weeks
  Biomarker of inflammation
interferon-alpha-21 | baseline and 2 weeks
  Biomarker of inflammation
interferon-gamma | baseline and 2 weeks
  Biomarker of inflammation
interleukin-1-alpha | baseline and 2 weeks
  Biomarker of inflammation
total cholesterol | baseline and 2 weeks
  lipid risk factor for cardiovascular disease
low-density lipoprotein-cholesterol | baseline and 2 weeks
  lipid risk factor for cardiovascular disease
high-density lipoprotein-cholesterol | baseline and 2 weeks
  lipid risk factor for cardiovascular disease
apolipoprotein-B | baseline and 2 weeks
  lipid risk factor for cardiovascular disease
fasting glucose | baseline and 2 weeks
  indicator of insulin resistance
systolic blood pressure | baseline and 2 weeks
  mmHg
diastolic blood pressure | baseline and 2 weeks
  mmHg
interleukin-6 | baseline and 2 weeks
  Biomarker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Sonia S Anand, MD, PhD, Principal Investigator — McMaster University; Hamilton Health Sciences Center; Population Health Research Institute
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Because sensitive genetic material was collected as part of this pilot study, data from this study will not be shared.

REFERENCES:
- [Background] Anand SS, Yusuf S. Stemming the global tsunami of cardiovascular disease. Lancet. 2011 Feb 12;377(9765):529-32. doi: 10.1016/S0140-6736(10)62346-X. Epub 2011 Feb 4. No abstract available. PMID 21295845
- [Background] O'Donnell CJ, Nabel EG. Genomics of cardiovascular disease. N Engl J Med. 2011 Dec 1;365(22):2098-109. doi: 10.1056/NEJMra1105239. No abstract available. PMID 22129254
- [Background] McPherson R, Pertsemlidis A, Kavaslar N, Stewart A, Roberts R, Cox DR, Hinds DA, Pennacchio LA, Tybjaerg-Hansen A, Folsom AR, Boerwinkle E, Hobbs HH, Cohen JC. A common allele on chromosome 9 associated with coronary heart disease. Science. 2007 Jun 8;316(5830):1488-91. doi: 10.1126/science.1142447. Epub 2007 May 3. PMID 17478681
- [Background] Do R, Xie C, Zhang X, Mannisto S, Harald K, Islam S, Bailey SD, Rangarajan S, McQueen MJ, Diaz R, Lisheng L, Wang X, Silander K, Peltonen L, Yusuf S, Salomaa V, Engert JC, Anand SS; INTERHEART investigators. The effect of chromosome 9p21 variants on cardiovascular disease may be modified by dietary intake: evidence from a case/control and a prospective study. PLoS Med. 2011 Oct;8(10):e1001106. doi: 10.1371/journal.pmed.1001106. Epub 2011 Oct 11. PMID 22022235
- [Background] Mente A, de Koning L, Shannon HS, Anand SS. A systematic review of the evidence supporting a causal link between dietary factors and coronary heart disease. Arch Intern Med. 2009 Apr 13;169(7):659-69. doi: 10.1001/archinternmed.2009.38. PMID 19364995
- [Background] Hu FB, Rimm EB, Stampfer MJ, Ascherio A, Spiegelman D, Willett WC. Prospective study of major dietary patterns and risk of coronary heart disease in men. Am J Clin Nutr. 2000 Oct;72(4):912-21. doi: 10.1093/ajcn/72.4.912. PMID 11010931